CLINICAL TRIAL: NCT04848259
Title: A Novel Therapeutic Approach for Controlling Complications Associated With Impacted Mandibular Third Molar Removal
Brief Title: Effect of Honey and Dexamethason on Extraction Healing
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Alaa Altaweel, Associate professor, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Impaction
Record Dates: First submitted 2021-04-14; First posted 2021-04-19 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Impacted Third Molar Tooth
MeSH Terms: interventions — Saline Solution; Dexamethasone; Honey

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control (Placebo Comparator): No drug given before surgery
  Interventions: Drug: Normal saline
- Dexamethason (Active Comparator): Dexamethason will be given IV before surgery
  Interventions: Drug: Dexamethasone
- Natural honey (Active Comparator): Honey will be placed locally after impaction removal
  Interventions: Drug: Honey
- Dexamethason and natural honey (Active Comparator): Dexamethason will be given IV before surgery and Honey will be placed locally after impaction removal
  Interventions: Drug: Dexamethasone and honey

INTERVENTIONS:
Drug: Normal saline — Saline will be applied after surgery
  Arms: Control
Drug: Dexamethasone — Dexamethason will be given IV before surgery
  Arms: Dexamethason
Drug: Honey — Honey will be applied locally after surgery
  Arms: Natural honey
Drug: Dexamethasone and honey — Dexamethason will be given IV before surgery and then Honey will be applied locally after surgery
  Arms: Dexamethason and natural honey

SUMMARY:
Natural honey and dexamethason will be given before impaction removal then postoperative complications will be evaluated

DETAILED DESCRIPTION:
Patient with impacted lower third molar will be selected to this study agording to agent applied preoperative. Group 1 will receive topical honey and Group 2 will receive IV dexamethason. After surgical removal of impacted tooth under local anesthesia postoperative pain mouth opening, and swelling will be evaluated

ELIGIBILITY:
Inclusion Criteria:

* impacted 3rd molar
* healthy patient No smoking

Exclusion Criteria:

* history of smoking Medical disease

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2021-06-20 (Actual); Study Completion 2021-06-27 (Actual)

PRIMARY OUTCOMES:
Interincisal distance | Preoperative
  Distance between upper and lower teeth will be measured in mm by ruler
Interincisal distance | I day postoperative
  Distance between upper and lower teeth will be measured in mm by ruler
Interincisal distance | 3rd day postoperative
  Distance between upper and lower teeth will be measured in mm by ruler
Interincisal distance | 7th day postoperative
  Distance between upper and lower teeth will be measured in mm by ruler
Edema | Preoperative
  Measured from angle of mandible to angle of mouth
Edema | 1day postoperative
  Measured from angle of mandible to angle of mouth
Edema | 2nd day postoperative
  Measured from angle of mandible to angle of mouth in mm by ruler
Edema | 3rd day postoperative
  Measured from angle of mandible to angle hof mouth in mm by ruler
Edema | 7th day postoperative
  Measured from angle of mandible to angle of mouth in mm by ruler

CONTACTS AND LOCATIONS:
Locations (1):
- Vision colleges, Jeddah, Saudi Arabia